CLINICAL TRIAL: NCT04505488
Title: Efficacy of the ASD Screening and Parent ENgagement (ASPEN) Intervention Program in Low-Resource Communities
Brief Title: Efficacy of the ASPEN Intervention Program in Low-Resource Communities
Acronym: ASPEN
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Collaborators: National Institute on Disability, Independent Living, and Rehabilitation Research (U.S. Federal Agency)
Responsible Party: Principal Investigator, Sandra B. Vanegas, Research Assistant Professor, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 90IFST0004
Record Dates: First submitted 2020-07-18; First posted 2020-08-10 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism; Parent-mediated intervention; Naturalistic developmental behavioral intervention; Low resource households
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The intervention group will receive a parent manual, a resource packet, and 12 weekly sessions delivered by the clinician and peer leader.
  Interventions: Behavioral: ASD Screening Parent ENgagement Intervention Program (ASPEN)
- Control Group (No Intervention): The control group will receive a parent manual and a resource packet. Four phone check-ins will be conducted across 12-14 weeks to address questions by the research team.

INTERVENTIONS:
Behavioral: ASD Screening Parent ENgagement Intervention Program (ASPEN) — The ASPEN intervention is based on naturalistic developmental behavioral intervention strategies to support the development of social communication and play skills and reduce challenging behavior.
  Other Names: ASPEN
  Arms: Intervention Group

SUMMARY:
The ASD Screening and Parent ENgagement (ASPEN) program is a culturally adapted, parent-mediated intervention program. The ASPEN program is tailored to address social communication and behavioral difficulties that young children with developmental delays may experience in early childhood. The ASPEN Program includes 12 sessions where parents are provided with psychoeducation about self-care, child development, and evidence-based strategies. Coaching is also provided to train parents on using evidence-based strategies within the home setting. The ASPEN program is delivered by a student clinician and a peer leader. We hypothesize that coaching strategies delivered by the clinician will lead to primary family caregivers learning evidence-based strategies and this will result in improved child outcomes. We hypothesize that education and family support delivered by peer leaders will help primary family caregivers learn social support strategies and this will lead to improved parent outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Child is between 18 months through 6 years of age
* Child has a medical diagnosis or educational classification of Autism or Autism Spectrum Disorder (ASD) or child is at-risk for Autism/ASD as determined by the Modified-Checklist for Autism in Toddlers - Revised/Follow-up Interview (M-CHAT-R/F) and/or Social Communication Questionnaire (SCQ)
* Child resides in a low-resource household as determined by at least one of the following criteria:
* -Child or family has Medicaid as an insurance provider
* -Child's primary caregiver has achieved a high school or lower education
* -Child resides in a household with an annual income of 200% of the Federal Poverty Level

Exclusion Criteria:

* Primary caregiver does not speak/understand English or Spanish
* Child is younger 18 months or older than 6 years of age
* Child does not have a medical diagnosis or educational classification of Autism/ASD or does not meet at-risk criteria on the M-CHAT-R/F and/or SCQ
* Child does not reside in low-resource household

Ages: 18 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 320 (Estimated)
Dates: Start 2020-07-07 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Adaptive Behavior | Baseline to Post-Intervention (12-14 weeks post baseline) Change
  Vineland Adaptive Behavior Scales - 3: Adaptive Behavior Composite Standard Score Minimum value = 20; Maximum value = 140; Higher scores indicate a better outcome
Adaptive Behavior | Baseline to Follow-Up (24-28 weeks post baseline) Change
  Vineland Adaptive Behavior Scales - 3: Adaptive Behavior Composite Standard Score Minimum value = 20; Maximum value = 140; Higher scores indicate a better outcome
Parenting Stress | Baseline to Post-Intervention (12-14 weeks post baseline) Change
  Parenting Stress Index - Short Form Total Stress T Score Minimum value = 32; Maximum value = 92; Higher scores indicate a worse outcome
Parenting Stress | Baseline to Follow-Up (24-28 weeks post baseline) Change
  Parenting Stress Index - Short Form Total Stress T Score Minimum value = 32; Maximum value = 92; Higher scores indicate a worse outcome
Parent Empowerment | Baseline to Post-Intervention (12-14 weeks post baseline) Change
  Family Outcomes Scales - Revised Minimum value = 1; Maximum value = 5; Higher scores indicate a better outcome
Parent Empowerment | Baseline to Follow-Up (24-28 weeks post baseline) Change
  Family Outcomes Scales - Revised Minimum value = 1; Maximum value = 5; Higher scores indicate a better outcome

SECONDARY OUTCOMES:
Child Challenging Behavior | Baseline to Post-Intervention (12-14 weeks post baseline) Change
  Scales of Independent Behavior-Revised: Problem Behavior Subscale Minimum value = +10; Maximum value = -74; Higher scores indicate a better outcome
Child Challenging Behavior | Baseline to Follow-Up (24-28 weeks post baseline) Change
  Minimum value = +10; Maximum value = -74; Higher scores indicate a better outcome
Family Quality of Life | Baseline to Post-Intervention (12-14 weeks post baseline) Change
  PedsQL Family Impact Module: Family Functioning Minimum value = 0; Maximum value = 100; Higher scores indicate a better outcome
Family Quality of Life | Baseline to Follow-Up (24-28 weeks post baseline) Change
  PedsQL Family Impact Module: Family Functioning Minimum value = 0; Maximum value = 100; Higher scores indicate a better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Sandra B Vanegas, PhD, Principal Investigator — University of Texas at Austin
Locations (1):
- University of Texas at Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: Data will be available 1 year after study completion.
Access Criteria: Electronic data from assessments will be submitted to Inter-university Consortium for Political and Social Research within 1 year after study completion for archival and storage purposes.